CLINICAL TRIAL: NCT00495625
Title: Phase II Open-Label Study of Sunitinib Malate (SUO11248) in Adult Subjects With Metastatic and/or Surgically Unresectable Hepatocellular Cancers (HCC)
Brief Title: Sunitinib Malate (SUO11248) In Subjects W/ Metastatic And/Or Surgically Unresectable Hepatocellular Cancers (HCC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-14733; Pfizer #2005-0880 (Other: Pfizer)
Record Dates: First submitted 2007-06-29; First posted 2007-07-03 (Estimated); Results first posted 2012-03-23 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2011-12

CONDITIONS: Liver Cancer
Keywords: Hepatocellular cancer (HCC); Sunitinib malate; Vascular endothelial growth factor (VEGF); Platelet-derived growth factor (PDGF); Tyrosine kinases; Liver
MeSH Terms: conditions — Liver Neoplasms | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sunitinib Malate (SUO11248) Treatment (Experimental)
  Interventions: Drug: Sunitinib Malate

INTERVENTIONS:
Drug: Sunitinib Malate — Once daily oral doses on days 1-28 of each 42-day cycle. The dose for the first 2 cycles will be 37.5 mg daily for 28 days, every 42 days. Dose may be escalated to 50 mg daily for 28 days at the treating investigator's discretion.
  Other Names: SU011248; Sutent

SUMMARY:
An open label multi-site phase II clinical trial of dose escalated sunitinib malate given orally once daily on days 1-28 of each 42-day cycle. Treatment will be continued until there is either disease progression or cumulative or acute toxicity which in the opinion of the treating physician compromises the ability of the patient to receive treatment or patient desire to stop treatment.

DETAILED DESCRIPTION:
An open label multi-site phase II clinical trial of sunitinib malate given orally once daily on days 1-28 of each 42-day cycle. Sunitinib malate will be dispensed as capsules at the beginning of each treatment cycle. The dose may be escalated at the investigator's discretion. Treatment will be continued until there is either disease progression or cumulative or acute toxicity which in the opinion of the treating physician compromises the ability of the patient to receive treatment or patient desire to stop treatment.

A follow up visit will be required before the beginning of every cycle every 6 weeks to assess toxicity and for physical examination. Complete blood count (CBC) and differential, comprehensive metabolic panel (including liver function tests) and alpha-feto protein (when indicated) will be obtained at every scheduled follow up visit.

ELIGIBILITY:
Inclusion Criteria:

* Resolution of all acute toxic effects of prior chemotherapy or radiotherapy or surgical procedures to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 grade less than or equal to 1.
* Adequate organ function as defined by the following criteria:

  * Serum aspartate transaminase (AST); serum glutamic oxaloacetic transaminase (SGOT) and serum alanine transaminase (ALT); serum glutamic pyruvic transaminase (SGPT) less than or equal to 2.5 x local laboratory upper limit of normal (ULN), or AST and ALT less than or equal to 5 x ULN if liver function abnormalities are due to underlying malignancy
  * Total serum bilirubin less than or equal to 1.5 x ULN
  * Absolute neutrophil count (ANC) more than or equal to 1500/mcL
  * Platelets more than or equal to 100,000/mcL
  * Hemoglobin more than or equal to 9.0 g/dL
  * Serum calcium less than or equal to 12.0 mg/dL
  * Serum creatinine less than or equal to 1.5 x ULN
* Biopsy-proven disease
* Measurable disease radiographically
* Disease that is deemed surgically unresectable (awaiting orthotopic hepatic transplantation allowable) and/or metastatic
* Age greater or equal to 18 years
* Life expectancy greater than 16 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2 (Karnofsky score > 60%)

Exclusion Criteria:

* Major surgery or radiation therapy or chemotherapy within 4 weeks of starting the study treatment
* NCI CTCAE version 3 grade 3 hemorrhage within 4 weeks of starting the study treatment
* History of or known brain metastases, spinal cord compression, or carcinomatous meningitis, or evidence of symptomatic brain or leptomeningeal disease on screening computed tomography (CT) or magnetic resonance imaging (MRI) scan
* Any of the following within the 6 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism.
* Known brain metastases
* Ongoing cardiac dysrhythmias of NCI CTCAE grade greater than or equal to 2
* Ongoing cardiac dysrhythmias of NCI CTCAE grade greater than or equal to 2, atrial fibrillation of any grade, or prolongation of the QTc interval to > 450msec for males or > 470 msec for females
* Hypertension that cannot be controlled by medications (>150/100 mm Hg despite optimal medical therapy)
* Pre-existing thyroid abnormality with thyroid function that cannot be maintained in the normal range with medication
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness or other active infection
* Concurrent treatment on another clinical trial; supportive care trials or non-treatment trials, e.g. Quality of Life (QOL), are allowed
* Concomitant use of ketoconazole or other agents known to induce CYP3A4
* Concomitant use of theophylline and phenobarbital and/or other agents metabolized by the cytochrome P450 system
* Ongoing treatment with therapeutic doses of Coumadin (low dose Coumadin up to 2 mg po daily for thrombo prophylaxis is allowed)
* Pregnancy or breastfeeding. Female subjects must be surgically sterile or be postmenopausal, or must agree to use effective contraception during the period of therapy. All female subjects with reproductive potential must have a negative pregnancy test (serum or urine) prior to enrollment. Male subjects must be surgically sterile or must agree to use effective contraception during the period of therapy. The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2006-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Strosberg, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: H Lee Moffitt Cancer Center & Research Institute website — http://www.moffitt.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients with unresectable or metastatic hepatocellular cancer (HCC) seen at the Moffitt Cancer Center Gastrointestinal (GI) Clinic were screened for eligibility to be enrolled in the study.
Groups:
- Sunitinib Malate (SUO11248) Treatment: Once daily oral doses on days 1-28 of each 42-day cycle. The dose for the first 2 cycles was 37.5 mg daily for 28 days, every 42 days. Dose could be escalated to 50 mg daily for 28 days at the treating investigator's discretion.
Period: Overall Study
Arm/Group | Sunitinib Malate (SUO11248) Treatment
Started | 33
Completed | 23
Not Completed | 10
Not completed — Did not complete at least 1 42 day cycle | 10

BASELINE CHARACTERISTICS:
Arm/Group | Sunitinib Malate (SUO11248) Treatment
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 12
Age Continuous [Mean (Full Range); unit: years] | 60.65 [24 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 26
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Partial Response (PR) at Interim Analysis
Description: Partial Response at Interim Analysis. Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (unidimensional measurement) of target lesions, taking as reference the baseline sum longest diameter (LD). Response was evaluated using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee [JNCI 92(3):205-216, 2000].
Time Frame: On Treatment to Off Study - average of 7 months per participant
Population: 17 of the 23 patients that were enrolled at time of Interim Analysis (patients enrolled between 10/13/06 and 9/24/07) were evaluable for response.
Measure: Number; unit: participants
Arm/Group | Sunitinib Malate (SUO11248) Treatment
Number analyzed (Participants) | 17
participants | 1

2. Secondary Outcome: Participant Time to Tumor Progression (TTP)
Description: Investigators planned to determine the time to tumor progression (TTP) of sunitinib malate in the treatment in unresectable Hepatocellular Cancers (HCC). TTP is defined as the duration of time from start of treatment to time of progression.
Time Frame: On Treatment to Off Study - average of 7 months per participant
Population: Not analyzed. The Principal Investigator who initiated the study left Moffitt before reaching the target enrollment required to perform the planned analysis.
Measure: Mean (Full Range); unit: months
Arm/Group | Sunitinib Malate (SUO11248) Treatment
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants With Overall Survival (OS)
Description: Overall survival (OS) of sunitinib malate in the treatment in unresectable HCC
Time Frame: On Treatment to Off Study - average of 7 months per participant
Population: Participants who had not expired on their off study date.
Measure: Number; unit: participants
Arm/Group | Sunitinib Malate (SUO11248) Treatment
Number analyzed (Participants) | 33
participants | 20

4. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: The toxicity of sunitinib malate in the treatment in unresectable HCC
Time Frame: On Treatment to Off Study - average of 7 months per participant
Population: All participants
Measure: Number; unit: participants
Arm/Group | Sunitinib Malate (SUO11248) Treatment
Number analyzed (Participants) | 33
participants | 11

5. Primary Outcome: Number of Participants With Stable Disease (SD) at Interim Analysis
Description: Stable Disease (SD) Rate at Interim Analysis. Stable Disease (SD): Neither sufficient shrinkage to qualify for Partial Response (PR) nor sufficient increase to qualify for Progressive Disease (PD), taking as reference the smallest sum longest diameter (LD) since the treatment started. Response and progression were evaluated in this study using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee [JNCI 92(3):205-216, 2000].
Time Frame: On Treatment to Off Study - average of 7 months per participant
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Sunitinib Malate (SUO11248) Treatment
Number analyzed (Participants) | 17
participants | 6

6. Primary Outcome: Number of Participants With Progressive Disease (PD) at Interim Analysis
Description: Progressive Disease Rate. Progressive Disease (PD): At least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Response and progression were evaluated in this study using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee [JNCI 92(3):205-216, 2000].
Time Frame: On Treatment to Off Study - average of 7 months per participant
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Sunitinib Malate (SUO11248) Treatment
Number analyzed (Participants) | 17
participants | 8

ADVERSE EVENTS:
Time Frame: 3 Years and 4 Months
Description: First Treatment Start Date: 10/13/06 Last Off Study Date: 2/19/10
Arm/Group | Sunitinib Malate (SUO11248) Treatment
Serious Adverse Events (participants affected / at risk) | 11/33
Other Adverse Events (participants affected / at risk) | 31/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sunitinib Malate (SUO11248) Treatment (N=33)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1) — Grade 3 - Unrelated
Death - Disease Progression (General disorders) | 4 (4) — Grade 5 - Death not associated with CTCAE term - Unrelated
Sudden Death (General disorders) | 1 (1) — Grade 5 - Death not associated with CTCAE term - unlikely that it is related
Ascites - Non-malignant (Gastrointestinal disorders) | 1 (1) — Grade 3 - Unrelated
Dehydration (Gastrointestinal disorders) | 1 (1) — Grade 3 - Probably related
Diarrhea (Gastrointestinal disorders) | 1 (1) — Grade 3 - Probably related
Nausea (Gastrointestinal disorders) | 1 (1) — Grade 3 - Probably related
Vomiting (Gastrointestinal disorders) | 1 (1) — Grade 3 - Probably related
Infection with normal ANC or Grade 1 or 2 neutrophils - Wound (Infections and infestations) | 1 (1) — Grade 3 - Unrelated
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 (1) — Grade 1 - Unrelated
Sodium, serum -low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1) — Grade 1 - Unrelated
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1) — Grade 3 - Unrelated
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 2 - Unrelated
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1) — Grade 2 - Unrelated
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sunitinib Malate (SUO11248) Treatment (N=33)
Diarrhea (Gastrointestinal disorders) | 15 (22)
Nausea (Gastrointestinal disorders) | 15 (18)
Anorexia (Gastrointestinal disorders) | 12 (13)
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 9 (11)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 8 (12)
Vomiting (Gastrointestinal disorders) | 7 (8)
Heartburn/dyspepsia (Gastrointestinal disorders) | 6 (6)
Gastrointestinal - Other (Gastrointestinal disorders) | 5 (7)
Dehydration (Gastrointestinal disorders) | 3 (3)
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 3 (3)
Ascites (non-malignant) (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Distension/bloating, abdominal (Gastrointestinal disorders) | 2 (2)
Flatulence (Gastrointestinal disorders) | 2 (3)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 19 (22)
Fever (General disorders) | 3 (3) — Fever (in the absence of neutropenia, where neutropenia is defined as ANC<1.0 x 10^9/L)
Insomnia (General disorders) | 3 (3)
Rigors/chills (General disorders) | 2 (2)
Weight loss (General disorders) | 2 (2)
Sweating (diaphoresis) (General disorders) | 1 (2)
Weight gain (General disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 9 (18)
Hemolysis (e.g., immune hemolytic anemia, drug-related hemolysis) (Blood and lymphatic system disorders) | 8 (15)
Platelets (Blood and lymphatic system disorders) | 7 (14)
Hemoglobin (Blood and lymphatic system disorders) | 4 (6)
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 2 (2)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 7 (9)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 6 (11)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 5 (6)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 3 (3)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 (5)
Constitutional symptoms - Other (General disorders) | 4 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 (1)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Pain - Abdomen NOS (General disorders) | 7 (9)
Pain - Head/headache (General disorders) | 5 (7)
Pain - Back (General disorders) | 3 (3)
Pain - Muscle (General disorders) | 3 (3)
Pain - Extremity-limb (General disorders) | 2 (3)
Pain - Bone (General disorders) | 1 (1)
Pain - Joint (General disorders) | 1 (1)
Pain - Oral-gums (General disorders) | 1 (1)
Paiin - Other (General disorders) | 1 (1)
Pain - Testicle (General disorders) | 1 (1)
Pain - Tumor (General disorders) | 1 (3)
Thrombotic microangiopathy (e.g., thrombotic thrombocytopenic purpura [TTP] or hemolytic uremic synd (Blood and lymphatic system disorders) | 10 (21)
Coagulation - Other (Blood and lymphatic system disorders) | 1 (1)
INR (International Normalized Ratio of prothrombin time) (Blood and lymphatic system disorders) | 1 (1)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 8 (8)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 4 (5)
ALT, SGPT(serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 3 (5)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2 (2)
Alkaline phosphatase (Metabolism and nutrition disorders) | 2 (2)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1 (1)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1 (1)
Mental status (Psychiatric disorders) | 2 (2)
Mood alteration - Depression (Psychiatric disorders) | 2 (2)
Cognitive disturbance (Psychiatric disorders) | 1 (1)
Dizziness (General disorders) | 1 (2)
Extrapyramidal/involuntary movement/restlessness (General disorders) | 1 (1)
Memory impairment (General disorders) | 1 (1)
Mood alteration - Anxiety (Psychiatric disorders) | 1 (1)
Neuropathy: motor (General disorders) | 1 (1)
Somnolence/depressed level of consciousness (General disorders) | 1 (1)
Syncope (fainting) (General disorders) | 1 (1)
Tremor (General disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Edema: limb (Blood and lymphatic system disorders) | 6 (6)
Edema: head and neck (Blood and lymphatic system disorders) | 1 (1)
Edema: trunk/genital (Blood and lymphatic system disorders) | 1 (1)
Renal/Genitourinary - Other (Renal and urinary disorders) | 2 (2)
Incontinence, urinary (Renal and urinary disorders) | 1 (1)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1 (1)
Urine color change (Renal and urinary disorders) | 1 (1)
Hypertension (Cardiac disorders) | 3 (3)
Thyroid function, high (hyperthyroidism, thyrotoxicosis) (Endocrine disorders) | 2 (2)
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 1 (1)
Febrile neutropenia (Infections and infestations) | 1 (1) — Fever of unknown origin without clinically or microbiologically documented infection ANC<1.0 x 10^9/L, fever >=38.5 degrees C
Infection with noral ANCl or lGrade 1 or 2 neutrophils - Urinary tract NOS (Infections and infestations) | 1 (1)
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) — Generalized or specific area (not due to neuropathy) - Extremity - lower
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) — Generalized or specific area (not due to neuropathy) - Whole body/generalized
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 1 (1)
Watery eye (epiphora, tearing) (Eye disorders) | 2 (2)
Phlebitis (including superficial thrombosis) (Vascular disorders) | 1 (1)
Supraventricular and nodal arrhythmia - Sinus tachycardia (Cardiac disorders) | 1 (1)
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (2)
Flu-like syndrome (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The Principal Investigator who initiated the study left Moffitt before reaching the target enrollment required to perform the planned analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No